CLINICAL TRIAL: NCT02224391
Title: Smartphone-Delivered Attentional Bias Modification Training for Quitting Smokers
Brief Title: Smartphone-Delivered Attentional Bias Modification Training in Helping Patients Quit Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-0999; NCI-2015-00609 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-0999 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Results first posted 2022-09-28 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Current Every Day Smoker
MeSH Terms: interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (ABM training) (Experimental): Patients receive ABM training over 30 minutes through a smartphone on days 1-14. Patients then receive nicotine patches for up to 8 weeks.
  Interventions: Behavioral: Computer-Assisted Smoking Cessation Intervention; Other: Laboratory Biomarker Analysis; Drug: Nicotine Patch; Other: Questionnaire Administration
- Arm II (sham training) (Sham Comparator): Patients undergo sham training on days 1-14. Patients then receive nicotine patches for up to 8 weeks.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Nicotine Patch; Other: Questionnaire Administration; Other: Sham Intervention

INTERVENTIONS:
Behavioral: Computer-Assisted Smoking Cessation Intervention — Receive ABM training via a smartphone
  Arms: Arm I (ABM training)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nicotine Patch — Given via transdermal patch
  Other Names: NicoDerm CQ; Nicotine Skin Patch; Nicotine Transdermal Patch
Other: Questionnaire Administration — Ancillary studies
Other: Sham Intervention — Undergo sham training
  Arms: Arm II (sham training)

SUMMARY:
This randomized clinical trial studies how well a smartphone-delivered attentional bias modification training works in helping patients quit smoking. Smartphone-delivered attentional bias modification training may help patients quit smoking by reducing the attentional bias (the tendency of one's perception to be affected by their recurring thoughts) towards smoking cues that developed over time as a result of conditioning processes through which smoking cues become important.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of smartphone-delivered, in-home attentional bias modification (ABM) to reduce attentional bias (AB) to smoking cues and to reduce smoking behavior in the short- and long-term.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive ABM training over 30 minutes through a smartphone on days 1-14. Patients then receive nicotine patches for up to 8 weeks.

ARM II: Patients undergo sham training on days 1-14. Patients then receive nicotine patches for up to 8 weeks.

After completion of study treatment, patients are followed up on days 15, 29, 43, 57, and 72.

ELIGIBILITY:
Inclusion Criteria:

* Smoke an average of 5 or more cigarettes or little cigars per day (CPD) prior to telephone screen
* Produce an expired carbon monoxide (CO) level greater than or equal to 6 parts per million (ppm) or a NicAlert reading of > 2
* Have a working telephone
* Interested in quitting smoking in the next 30 days
* Fluency in spoken and written English
* Must sign the picture consent form

Exclusion Criteria:

* Taking psychotropic, anticonvulsive, or narcotic medication
* Meet criteria for a current major depressive episode or suicidality
* Have a history of neurological illness or closed head injury
* Report uncorrected vision problems
* Involved in current smoking cessation activity
* Testing positive on a urine drug screen for drugs of abuse/potential abuse
* Women who are pregnant or breastfeeding
* Considered by the investigator to be an unsuitable or unstable candidate (e.g., due to cognitive impairment)
* Shares the same address as a currently enrolled participant
* Unwilling to alter or remove hairstyle, hair extensions, or wig during the clinic visits to allow for correct electroencephalography (EEG) sensor placement
* Reports diagnosis of seizure disorder
* Unwilling to use nicotine replacement therapy (NRT) patches

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Robinson, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Robinson JD, Cui Y, Engelmann JM, Kypriotakis G, Cinciripini PM. Using eye tracking to evaluate the impact of smartphone-delivered attentional bias modification training for smokers. Exp Clin Psychopharmacol. 2024 Dec;32(6):728-736. doi: 10.1037/pha0000729. Epub 2024 Jun 27. PMID 38934914
- [Derived] Robinson JD, Cui Y, Linares Abrego P, Engelmann JM, Prokhorov AV, Vidrine DJ, Shete S, Cinciripini PM. Sustained reduction of attentional bias to smoking cues by smartphone-delivered attentional bias modification training for smokers. Psychol Addict Behav. 2022 Nov;36(7):906-919. doi: 10.1037/adb0000805. Epub 2022 Jan 13. PMID 35025555
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 246 participants were randomized
Groups:
- Arm I: Attention Bias Modification (ABM) Training: Patients receive ABM training over 30 minutes through a smartphone on days 1-14. Patients then receive nicotine patches for up to 8 weeks.
- Arm II: Sham Training: Patients undergo sham training on days 1-14. Patients then receive nicotine patches for up to 8 weeks.
Period: Overall Study
Arm/Group | Arm I: Attention Bias Modification (ABM) Training | Arm II: Sham Training
Started | 124 | 122
Completed | 92 | 98
Not Completed | 32 | 24
Not completed — Lost to Follow-up | 26 | 19
Not completed — Withdrawal by Subject | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Attention Bias Modification (ABM) Training | Arm II: Sham Training | Total
Number analyzed (Participants) | 124 | 122 | 246
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.27 (10.13) | 45.28 (11.65) | 46.28 (10.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 44 | 89
  Male | 79 | 78 | 157
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 14 | 29
  Not Hispanic or Latino | 108 | 108 | 216
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 22 | 56
  White | 80 | 92 | 172
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 124 | 122 | 246
Years of education [Mean (Standard Deviation); unit: years] | 13.35 (1.86) | 13.72 (2) | 13.53 (1.94)
Number of Participants Employed [Count of Participants; unit: Participants] | 83 | 96 | 179
Fagerström Test for Nicotine Dependence (FTND) total score [Mean (Standard Deviation); unit: score on a scale] — The Fagerström Test for Nicotine Dependence (FTND), yes/no items are scored from 0 to 1 and multiple-choice items are scored from 0 to 3. The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the patient's physical dependence on nicotine.
  score on a scale | 4.82 (2.14) | 4.96 (2.11) | 4.89 (2.12)
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] | 18.14 (8.87) | 18.48 (9.27) | 18.31 (9.05)

OUTCOME MEASURES:

1. Primary Outcome: Modified Dot-probe Task
Description: Modified dot-probe task evaluated by using 2 (group: ABM vs. sham) X 3 (session: baseline, 1-day post-training, and 8-weeks post-training) linear mixed model using RT difference scores (neutral-cigarette) as the dependent measures and subject as the random effect.
Time Frame: Up to 8 weeks post-training
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | Arm I: Attention Bias Modification (ABM) Training | Arm II: Sham Training
Number analyzed (Participants) | 124 | 122
milliseconds
  Baseline | 5.49 (0.99) | 7.49 (1)
  1-day post-training | 2.42 (1.04) | 9.85 (1.03)
  8-weeks post-training | 4.94 (1.19) | 9.48 (1.14)

2. Primary Outcome: Smoking Stroop Task
Description: The Stroop task will consist of three blocks, with a 5-s rest period between blocks: (a) practice (40 trials), (b) neutral words (80 trials), and (c) smoking words (80 trials). The score will be calculated by taking the mean RT difference between the smoking and neutral words on trials with correct responses within the response window.
Time Frame: Up to 8 weeks post-training
Measure: Least Squares Mean (Standard Error); unit: milisecond
Arm/Group | Arm I: Attention Bias Modification (ABM) Training | Arm II: Sham Training
Number analyzed (Participants) | 124 | 122
milisecond
  Baseline | -6.57 (4.11) | 4.94 (4.15)
  1-day post-training | -2.38 (4.31) | 3.73 (4.29)
  8-weeks post-training | -4.59 (4.94) | 10.97 (4.7)

3. Secondary Outcome: Cigarette Per Day (CPD)
Description: Mean number of cigarettes per day smoked for the seven days preceding each time point.
Time Frame: Up to 8 weeks post-training
Measure: Least Squares Mean (Standard Error); unit: number of cigerettes
Arm/Group | Arm I: Attention Bias Modification (ABM) Training | Arm II: Sham Training
Number analyzed (Participants) | 124 | 122
number of cigerettes
  Baseline | 18.1 (0.8) | 18.45 (0.81)
  1-day post-training | 14.94 (0.82) | 14.78 (0.83)
  8-weeks post-training | 8.29 (0.9) | 7.52 (0.87)

4. Secondary Outcome: Expired Carbon Monoxide (CO)
Description: Mean expired carbon monoxide, in ppm (parts per million), at each time point.
Time Frame: Up to 8 weeks post-training
Measure: Least Squares Mean (Standard Error); unit: Parts Per Million
Arm/Group | Arm I: Attention Bias Modification (ABM) Training | Arm II: Sham Training
Number analyzed (Participants) | 124 | 122
Parts Per Million
  Baseline | 22.41 (1.1) | 22.27 (1.11)
  1-day post-training | 22.28 (1.13) | 22.95 (1.13)
  8-day post-training | 12.54 (1.24) | 12.99 (1.19)

5. Secondary Outcome: Urinary Cotinine
Description: Mean urinary cotinine, measured in ng/mL, at each time point.
Time Frame: Up to 8 weeks post-training
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Arm I: Attention Bias Modification (ABM) Training | Arm II: Sham Training
Number analyzed (Participants) | 124 | 122
ng/mL
  Baseline | 7.11 (.99) | 7.12 (.09)
  1-Day post-training | 6.91 (.09) | 6.99 (.09)
  8-Day post-training | 6.16 (.12) | 6.61 (.12)

6. Secondary Outcome: Fagerström Test for Nicotine Dependence (FTND)
Description: The Fagerström Test for Nicotine Dependence, yes/no items are scored from 0 to 1 and multiple-choice items are scored from 0 to 3. The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the patient's physical dependence on nicotine. Mean Fagerström Test for Nicotine Dependence (FTND) questionnaire score at each time point.
Time Frame: Up to 8 weeks post-training
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Arm I: Attention Bias Modification (ABM) Training | Arm II: Sham Training
Number analyzed (Participants) | 124 | 122
score on a scale
  Baseline | 4.84 (0.19) | 4.96 (0.19)
  1-day post-training | 4.34 (0.2) | 4.05 (0.2)
  8-weeks post-training | 2.93 (0.21) | 2.65 (0.21)

7. Secondary Outcome: Wisconsin Smoking Withdrawal Scale (WSWS) - Craving
Description: Mean Wisconsin Smoking Withdrawal Scale (WSWS) - Craving subscale score at each time point. Participants rate each item on a scale of 0-4 (0=Strongly disagree, 1=Disagree, 2=Feel neutral, 3=Agree, 4=Strongly agree). The subscale to each item is determined on how high they agree on the scale. Mean Wisconsin Smoking Withdrawal Scale (WSWS) - Craving subscale score at each time point. For some items, the subscale is determined on how low they agreed. Each score is determined by the mean of each item that applies. Higher means indicate greater withdrawal.
Time Frame: Up to 8 weeks post-training
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Arm I: Attention Bias Modification (ABM) Training | Arm II: Sham Training
Number analyzed (Participants) | 124 | 122
score on a scale
  Baseline | 9.9 (0.29) | 9.76 (0.29)
  1-day post-training | 8.36 (0.3) | 8.52 (0.3)
  8-weeks post-training | 6.92 (0.34) | 6.73 (0.32)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Per the trial only adverse events potentially related to use of the nicotine patch were reported. Internal Serious Adverse Events (SAE) that are unexpected (not listed in the Informed Consent Document) and are related (possible, probable and definite) must be reported to the IRB within 5 working days. Deaths that are related and occur within 30 days after completion of treatment must be submitted to the IRB within 24 hours.
Arm/Group | Arm I: Attention Bias Modification (ABM) Training | Arm II: Sham Training
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/122
Serious Adverse Events (participants affected / at risk) | 4/124 | 2/122
Other Adverse Events (participants affected / at risk) | 60/124 | 67/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Attention Bias Modification (ABM) Training (N=124) | Arm II: Sham Training (N=122)
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Attention Bias Modification (ABM) Training (N=124) | Arm II: Sham Training (N=122)
Abnormal dreams (Nervous system disorders) | 19 | 19
Anxiety (Psychiatric disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Concentration impairment (Nervous system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2
Dizziness (Nervous system disorders) | 5 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 5 | 5
Insomnia (Psychiatric disorders) | 15 | 10
Irritability (Psychiatric disorders) | 0 | 1
Mucosal infection (Infections and infestations) | 2 | 0
Nausea (Gastrointestinal disorders) | 5 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 32 | 42
Stomach pain (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT02224391/Prot_SAP_000.pdf